CLINICAL TRIAL: NCT06875583
Title: The Radiation ProtEction for Dose RedUction in the Cardiac CathEter Lab Study: The REDUCE Trial
Acronym: REDUCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Rampart Health, L.L.C. (Industry)
Responsible Party: Principal Investigator, John Hung, Consultant Cardiologist, Chief Investigator, Liverpool Heart and Chest Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REDUCE
Record Dates: First submitted 2025-02-17; First posted 2025-03-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Radiation Exposure; Radiation Exposure to Operator; Radiation Injuries; Radiation Safety
Keywords: radiation exposure; radiation exposure to operator; radiation injuries; radiation safety
MeSH Terms: conditions — Radiation Injuries | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Multi-centre randomised controlled trial. Coronary catheter laboratory procedures will be randomised 1:1 to RAMPART vs standard radiation protection using a pre-defined randomisation schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAMPART Arm (Experimental): The use of the RAMPART system to reduce operator radiation exposure
  Interventions: Device: Radiation
- Standard Arm (No Intervention): Standard radiation protection

INTERVENTIONS:
Device: Radiation — The use of RAMPART radiation protection device
  Other Names: Use of RAMPART radiation protection device
  Arms: RAMPART Arm

SUMMARY:
Doctors and nurses who perform heart procedures using X-ray guidance are exposed to radiation, which can be harmful over time. This exposure increases the risk of certain health problems, including cancers, eye damage (cataracts), and DNA damage. Although protective lead clothing is used to reduce exposure, it is heavy, uncomfortable, and can cause muscle and joint problems for those who wear it daily.

A new radiation protection device, called RAMPART, may help reduce radiation exposure for heart specialists and their teams. It could also allow them to wear lighter protective gear-or none at all-making their work safer and more comfortable.

This study will compare the radiation levels received by doctors and nurses during heart procedures when using RAMPART versus standard protection. By doing so, we hope to find out if this new device can better protect medical teams from radiation, improving both their safety and well-being.

DETAILED DESCRIPTION:
Recent decades have seen major increases in x-ray guided procedures in interventional cardiology, radiology and vascular surgery. Exposure to ionising radiation is known to be an inherent risk and remains a serious and unresolved threat to the health of operators and their team. It is associated with an increased incidence of brain and blood cancers, cataracts, and recent mechanistic data indicates significantly increased DNA damage in those without leaded leg protection.

Although existing standard radiation protection measures somewhat reduces exposure, all cardiac catheter lab personnel still receive a certain dose of radiation and continue to accumulate lifetime exposure. Furthermore, leaded personal protective equipment is heavy, leads to orthopaedic complications, and detracts from operator comfort.

Novel radiation protection devices such as RAMPART may significantly reduce radiation doses to cardiac catheter lab personnel, and potentially allow the use of lighter lead, or no lead at all. In this study we aim to investigate if use of RAMPART significantly reduces radiation exposure, when compared with standard radiation protection. Standard coronary intervention procedures will be randomised to RAMPART or standard (radiation protection), and operators and Cath lab team doses will be compared.

ELIGIBILITY:
Inclusion Criteria:

* All procedures involving adult patients (>18 year of age)
* Male or female patients
* Planned to undergo either an elective or urgent coronary intervention procedure involving ionising radiation in the cardiac catheter lab, via the right and or left radial arteries.

Exclusion Criteria:

* Procedures involving patients less than 18 years of age
* Patients unable to give valid consent
* Pregnancy
* Femoral approach procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
1st Operator Eye radiation | 1) Periprocedural 2) Cumulative dose - through study completion, an average of 1 year
  To assess the effect of using a new medical device (RAMPART) in reducing the amount of radiation the first operator is exposed to (at eye level) when performing coronary angiography or angioplasty. Measurement of radiation in µSv.

SECONDARY OUTCOMES:
1st Operator Chest / Groind radiation | 1) Periprocedural 2) Cumulative dose - through study completion, an average of 1 year
  To assess if RAMPART significantly reduces the radiation dose to first operators during coronary angiography or angioplasty at chest and groin level. Measurement of radiation in µSv.
2nd Operator Radiation - all levels | 1) Periprocedural 2) Cumulative dose - through study completion, an average of 1 year
  To assess if RAMPART significantly reduces the radiation dose to second operators during coronary angiography or angioplasty at the level of eye, chest and groin. Measurement of radiation in µSv.
'Circulating Nurse' Radiation | 1) Periprocedural 2) Cumulative dose - through study completion, an average of 1 year
  To assess if RAMPART significantly reduces radiation dose in a more distant position, consistent with that of a 'circulating nurse'. Measurement of radiation in µSv.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool Heart & Chest Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Direct access will be granted to the Sponsor, host institution and the regulatory authorities to permit trial-related monitoring, audits and inspections in line with participant consent. Furthermore, all data will be shared through publication and via online additional data supplements.
Supporting Information: Study Protocol, CSR
Time Frame: End of trial and publication
Access Criteria: 1. Published Journal platform
  2. Open Source Framework - https://osf.io/
URL: https://osf.io/

REFERENCES:
- [Result] Lisko JC, Shekiladze N, Chamoun J, Sheikh N, Rainer K, Wei J, Binongo J, Raj L, Byku I, Rinfret S, Devireddy C, Jaber WA, Greenbaum AB, Babaliaros V, Steuterman S, Sandesara P, Nicholson WJ. Radiation Exposure Using Rampart vs Standard Lead Aprons and Shields During Invasive Cardiovascular Procedures. J Soc Cardiovasc Angiogr Interv. 2023 Oct 19;3(1):101184. doi: 10.1016/j.jscai.2023.101184. eCollection 2024 Jan. PMID 39131978
- [Result] Noor HA, Althawadi N, Noor Z, AlAnsari N, Chachar TS, Al Raisi S, Yousif N. Radiation Exposure During Invasive Cardiovascular Procedures: Portable Shielding System Versus Standard Lead Aprons. Cureus. 2024 Aug 29;16(8):e68108. doi: 10.7759/cureus.68108. eCollection 2024 Aug. PMID 39350833